CLINICAL TRIAL: NCT05861570
Title: Steroid and Sodium Hyaluronate Hydrodilatation
Brief Title: Is Combined Steroid and Sodium Hyaluronate Hydrodilatation More Effective Than Isolated Steroid Hydrodilatation in Treating Patients With Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-01-001B
Record Dates: First submitted 2023-04-05; First posted 2023-05-17 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-04

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Saline Solution; Hyaluronic Acid; Lidocaine; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydrodilatation with steroid (Experimental): patient received ultrasound-guided 3cc NS + 40mg triamcinolone + 4cc xylocaine
  Interventions: Drug: normal saline; Drug: lidocaine hydrochloride; Drug: Triamcinolone Acetonide
- hydrodilatation with hyaluronic acid and steroid (Active Comparator): patient received ultrasound-guided 3cc hyaluronic acid + 40mg triamcinolone + 4cc xylocaine
  Interventions: Drug: (Sodium Hyaluronate (Hyruan One , LG); Drug: lidocaine hydrochloride; Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: normal saline — Ultrasound guided injection using 3ml normal saline
  Arms: hydrodilatation with steroid
Drug: (Sodium Hyaluronate (Hyruan One , LG) — Ultrasound guided injection using 3ml of Sodium Hyaluronate
  Arms: hydrodilatation with hyaluronic acid and steroid
Drug: lidocaine hydrochloride — Ultrasound guided injection using 4ml of 2% lidocaine hydrochloride (Xylocaine)
Drug: Triamcinolone Acetonide — ultrasound guided steroid injection using 4ml of 40mg triamcinolone acetonide

SUMMARY:
This study was conducted to compare the efficacy of hydrodilatation with steroid with hyaluronic acid and steroid for treating adhesive capsulitis.

DETAILED DESCRIPTION:
Design: a prospective, double-blinded, randomized, clinical trial

Patient and methods:

Patients with adhesive capsulitis for at least 3 months were enrolled and randomly allocated into group 1 (hydrodilatation with steroid ) and group 2 (hydrodilatation with hyaluronic acid and steroid). The patients were evaluated before treatment and were reevaluated 0, 6, and 12 weeks after the beginning of the treatment. Outcomes measures included a pain scale (visual analog scale), range of motion, Shoulder Pain And Disability Index

ELIGIBILITY:
Inclusion Criteria:

1. age 35-65 years
2. onset of shoulder stiffness since over a month
3. limitation in the passive range of motion (ROM) over 30° when compared with the contralateral side in at least two of these three movements: forward flexion, abduction, or external rotation.

Exclusion Criteria:

1. ultrasound findings of rotator cuff tears,
2. plain radiography findings of significant glenohumeral joint arthritis,
3. accompanying cervical radiculopathy,
4. systemic inflammatory joint disease,
5. intraarticular injection into the glenohumeral joint within the past 3 months
6. history of surgery on the affected shoulders,
7. regular use of systemic non-steroidal anti-inflammatory drugs or corticosteroids,
8. allergy to corticosteroid or lidocaine.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-04-06 (Estimated); Study Completion 2024-04-06 (Estimated)

PRIMARY OUTCOMES:
change in pain intensity | 0, 6, 12weeks
  pain intensity was measured by visual analog scale (0-10)

SECONDARY OUTCOMES:
change in Shoulder Pain And disability index | 0, 6, 12 weeks
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
change in glenohumeral joint range of motion | 0, 6, 12weeks
  Shoulder flexion, abduction, external rotation and internal rotation were measured with goniometer with patient in supine position.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan